CLINICAL TRIAL: NCT06602687
Title: Sperm Hyaluronic Binding Selection (PICSI): Impact on Embryo Aneuploid Status in Assisted Human Reproduction
Brief Title: PICSI Impact on Euploidy in Assisted Reproduction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Merrion Fertility Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MFC3
Record Dates: First submitted 2024-08-01; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Infertility
Keywords: PICSI; Sperm; Aneuploidy
MeSH Terms: conditions — Infertility; Aneuploidy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard ICSI (No Intervention): ICSI performed using standard sperm selection methods.
- PICSI (Experimental): ICSI performed using sperm selected based on hyaluronan binding (PICSI® dish, Cooper Surgical).
  Interventions: Device: PICSI

INTERVENTIONS:
Device: PICSI — The PICSI® dish is a CE marked medical device containing dots of a HA hydrogel (Cooper Surgical).
  Arms: PICSI

SUMMARY:
Hyaluronic acid (HA) is a major component of the cumulus complex surrounding oocytes. Intracytoplasmic sperm injection (ICSI) involves injection of a selected sperm into the oocyte. Embryologists select sperm with normal morphology and progressive motility. Physiologic intracytoplasmic sperm injection (PICSI) involves sperm selection for ICSI based on hyaluronan binding. Mature sperm which bind to HA have greater genomic integrity and reduced levels of DNA fragmentation. Earlier observational studies demonstrated improved outcomes in assisted reproductive technologies (ART) including improved clinical pregnancy rates, decreased miscarriage rates and higher live birth rates. A large multicentre randomized trial, the HABSelect trial, which included over 2,500 couples, found that PICSI did not improve term (>37 weeks gestation) live birth rates compared to standard ICSI. However, mechanistic analysis of the data from the HABSelect trial showed a significant reduction in miscarriage rates, most notable in couples where the woman was aged over 37 years where a significant reduction in miscarriage rate was seen (40% with ICSI vs 15% with PICSI). A 2021 retrospective sibling oocyte study, including 45 cycles, compared fertilisation and embryo development and found higher fertilisation rate in PICSI cycles. No difference was observed in clinical pregnancy rates; miscarriage rates and live birth rates were not reported. We aim to prospectively study PICSI vs standard ICSI in sibling oocytes to investigate if PICSI improves embryological and ART outcomes, particularly fertilisation rate, embryo euploid status and miscarriage rate, where the female patient is aged over 35 years.

ELIGIBILITY:
Inclusion Criteria:

* Couples undergoing a planned ICSI-PGT-A cycle using their own fresh gametes
* Female age > 35 years and/or Male age > 40 years
* Minimum of two mature eggs at time of egg maturity assessment

Exclusion Criteria:

* Couples undergoing a planned IVF cycle (even if converted to ICSI)
* Patients using donor gametes for an ICSI cycle
* Patients using frozen gametes for an ICSI cycle

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Euploidy rates | 4 weeks
  Primary outcome is rate of euploid embryos per cycle after preimplantation genetic testing for aneuploidy (PGT-A)

SECONDARY OUTCOMES:
Fertilisation rates | 24-48 hours
  Defined as number of 2PNs per oocyte injected
Blastocyst development and rate | 5 and 6 days
  Assessed on day 5 and day 6 according to Gardner grading system.
Positive hCG rate | 6-7 weeks
  Defined as detection of urinary human chorionic gonadotropin (hCG) per embryo transfer cycles.
Clinical pregnancy rate | 6-7 weeks
  Defined as number of fetal heartbeats/ gestational sacs identified by ultrasonographic visualisation at 6-7 weeks gestation per cycles started, oocyte retrievals or embryo transfer cycles.
Miscarriage rate | up to 22 weeks
  Defined as number of spontaneous losses of an intra-uterine pregnancy prior to 22 completed weeks of gestational age per embryo transfer cycles.
Live birth rate | 37-42 weeks
  Defined as number of live births at ≥37 weeks gestation per embryo transfer cycles

CONTACTS AND LOCATIONS:
Overall Officials: David Crosby, MD, Study Director — Merrion Fertility Clinic and the National Maternity Hospital
Locations (1):
- Merrion Fertility Clinic, Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No